CLINICAL TRIAL: NCT04708561
Title: Therapy of Non-literal Language Comprehension Disorders in Brain-damaged Individuals: Case Studies
Brief Title: Therapy of Pragmatic Disorders in Brain-damaged Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Neuchatel (Other)
Responsible Party: Principal Investigator, Marion Fossard, Professor, University of Neuchatel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Unine2020-00301
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Brain Injuries, Traumatic; Right Hemispheric Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Speech Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain-injured participants (Experimental)
  Interventions: Behavioral: Speech and language therapy

INTERVENTIONS:
Behavioral: Speech and language therapy — The intervention focuses on understanding the thoughts of the characters. Twenty written stories will be used, which end with statements that can be interpreted literally, ironically, as a lie, a request or a faux-pas (maladroitness). At the end of each story, the participant should explain what the characters want to mean by their statement.
  To help the participant in his understanding of the character's intention, he will be asked:
  1) To mention as many intentions as possible that can be associated with the target statement presented out of context (eg: "it's hot here" that can be interpreted literally, ironically, as a lie or a request) and to imagine contexts in connection with interpretation; 2. Analyze the relevant elements of the context (environment, the relationship between the characters, knowledge of the characters); 3. To judge the probability of the possible interpretations (pt 1) by justifying using the elements of the context analyzed previously (pt 2).

SUMMARY:
This study aims to assess speech therapy's effectiveness in understanding other people's thoughts (implied) using written stories. The main objective is to examine whether the therapy improves understanding of the stories worked on in the sessions. We also explore whether the observed progress is maintained one month after the end of treatment and whether it is generalized to neuropsychological tests, video material, and the participants' daily lives.

This therapy will be administered to four individuals with brain lesions, for six weeks, at the rate of two weekly sessions of one hour.

ELIGIBILITY:
Inclusion Criteria:

* Have been the victim, in adulthood, of a moderate to severe traumatic brain injury (TBI) or a stroke, with at least right frontal lesions (objectified by imaging). The time between the TBI or stroke and participation in this study should be greater than six months.
* Be of French mother tongue or have an excellent mastery of French.
* Be between 20 and 65 years old.
* Be right-handed
* Present problems in the understanding of non-literal language (irony, indirect requests), objectified by a neuropsychological examination.

Exclusion Criteria:

* Have a history of psychiatric disorder affecting social cognition (according to DSM-V criteria), and more specifically: autism, schizophrenia, bipolar disorders, major depressive disorders, borderline personality disorders, generalized anxiety disorders, obsessive-compulsive disorders, phobia social and eating disorders (anorexia, bulimia).
* Have chronic symptoms of an alcohol or drug dependence disorder (according to DSM-V criteria).
* Have significant uncorrected vision and/or hearing problems.
* Have aphasia and/or significant reading and comprehension problems.
* Present significant spatial neglect.
* Present an impaired capacity for judgment and discernment, objectified by a neuropsychological evaluation.
* Have been the victim of several TBI or stroke

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change from the score on the written task of comprehension of non-literal language 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  The non-literal language comprehension task includes written stories ending with a character's utterance that can be interpreted literally (e.g., "I'm mad at you" to signify her nervousness); ironically (e.g. "it was a fantastic play" to mean the play was bad); as an indirect request (e.g., "Caramels look good" to ask for a caramel); like a lie (e.g. "it was very nice"); like a faux-pas (e.g., criticizing a person without knowing that he or she hears everything).
  Following these stories, the participant must answer the question: "What does the character mean? ". Each story is scored 0-1-2 depending on the accuracy of the answer. The total score is thus obtained by adding the points received for each of the questions in the task's stories.
  The stories will be administered twice before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from the score on the written task of comprehension of non-literal language 1 month after the end of the therapy | Baselines, 1 month-follow-up
  The non-literal language comprehension task includes written stories ending with a character's utterance that can be interpreted literally (e.g., "I'm mad at you" to signify her nervousness); ironically (e.g. "it was a fantastic play" to mean the play was bad); as an indirect request (e.g., "Caramels look good" to ask for a caramel); like a lie (e.g. "it was very nice"); like a faux-pas (e.g., criticizing a person without knowing that he or she hears everything).
  Following these stories, the participant must answer the question: "What does the character mean? ". Each story is scored 0-1-2 depending on the accuracy of the answer. The total score is thus obtained by adding the points received for each of the questions in the task's stories.
  The stories will be administered twice before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from the score on the written task of comprehension of non-literal language 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  The non-literal language comprehension task includes written stories ending with a character's utterance that can be interpreted literally (e.g., "I'm mad at you" to signify her nervousness); ironically (e.g. "it was a fantastic play" to mean the play was bad); as an indirect request (e.g., "Caramels look good" to ask for a caramel); like a lie (e.g. "it was very nice"); like a faux-pas (e.g., criticizing a person without knowing that he or she hears everything).
  Following these stories, the participant must answer the question: "What does the character mean? ". Each story is scored 0-1-2 depending on the accuracy of the answer. The total score is thus obtained by adding the points received for each of the questions in the task's stories.
  The stories will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.

SECONDARY OUTCOMES:
Change from a nonverbal test of theory of mind 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  The nonverbal test of theory of mind (Sarfati et al., 1997) consists of choosing among 3 images (i.e., 3 intentions) the one that correctly ends the story.
  The test will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a nonverbal test of theory of mind 1 month after the end of the therapy | Baselines, 1 month-follow-up
  The nonverbal test of theory of mind (Sarfati et al., 1997) consists of choosing among 3 images (i.e., 3 intentions) the one that correctly ends the story.
  The test will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a nonverbal test of theory of mind 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  The nonverbal test of theory of mind (Sarfati et al., 1997) consists of choosing among 3 images (i.e., 3 intentions) the one that correctly ends the story.
  The test will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.
Change from a verbal test of theory of mind 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  The verbal test of theory of mind (TOM-15; Desgranges et al., 2012) consists of reading a story and then answering a question about a character's false belief
  The test will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a verbal test of theory of mind 1 month after the end of the therapy | Baselines, 1 month-follow-up
  The verbal test of theory of mind (TOM-15; Desgranges et al., 2012) consists of reading a story and then answering a question about a character's false belief
  The test will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a verbal test of theory of mind 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  The verbal test of theory of mind (TOM-15; Desgranges et al., 2012) consists of reading a story and then answering a question about a character's false belief
  The test will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.
Change from a test of inhibitory control 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  The test of inhibitory control (Hayling, Rouleau, 1998) consists in completing oral sentences with a word that is not semantically related.
  The test will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a test of inhibitory control 1 month after the end of the therapy | Baselines, 1 month-follow-up
  The test of inhibitory control (Hayling, Rouleau, 1998) consists in completing oral sentences with a word that is not semantically related.
  The test will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a test of inhibitory control 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  The test of inhibitory control (Hayling, Rouleau, 1998) consists in completing oral sentences with a word that is not semantically related.
  The test will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.
Change from a test of cognitive flexibility 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  The test of inhibitory control (TrailMaking Test, Reitan & Wolfson, 1993) consists of connecting by alternating numbers and letters in ascending and alphabetical order.
  The test will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a test of cognitive flexibility 1 month after the end of the therapy | Baselines, 1 month-follow-up
  The test of inhibitory control (TrailMaking Test, Reitan & Wolfson, 1993) consists of connecting by alternating numbers and letters in ascending and alphabetical order.
  The test will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a test of cognitive flexibility 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  The test of inhibitory control (TrailMaking Test, Reitan & Wolfson, 1993) consists of connecting by alternating numbers and letters in ascending and alphabetical order.
  The test will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.
Change from a test of working memory 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  In this test (PASAT, Gronwall, 1977), the participant hears numbers and must add each new number heard to the previous one.
  The test will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a test of working memory 1 month after the end of the therapy | Baselines, 1 month-follow-up
  In this test (PASAT, Gronwall, 1977), the participant hears numbers and must add each new number heard to the previous one.
  The test will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a test of working memory 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  In this test (PASAT, Gronwall, 1977), the participant hears numbers and must add each new number heard to the previous one.
  The test will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.
Change from a video task of non-literal language comprehension 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  This task includes 16 videos from TV shows. After each excerpt, the participant must explain what the actor wanted to mean by his statement.
  The task will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a video task of non-literal language comprehension 1 month after the end of the therapy | Baselines, 1 month-follow-up
  This task includes 16 videos from TV shows. After each excerpt, the participant must explain what the actor wanted to mean by his statement.
  The task will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a video task of non-literal language comprehension 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  This task includes 16 videos from TV shows. After each excerpt, the participant must explain what the actor wanted to mean by his statement.
  The test task will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.
Change from a daily life impact self-questionnaire 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  The ERF-CS (Echelle de Répercussion Fonctionnelle des troubles de la Cognition Sociale; Peyroux & Franck, 2014), administered to the participant, comprises 14 questions assessing four domains of social cognition: theory of mind, emotional processes, attributional style and social knowledge. The score range from 28 to 140 points. The higher the score, the greater the impact of the disorders is considered.
  The questionnaire will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a daily life impact self-questionnaire 1 month after the end of the therapy | Baselines, 1 month-follow-up
  The ERF-CS (Echelle de Répercussion Fonctionnelle des troubles de la Cognition Sociale; Peyroux & Franck, 2014), administered to the participant, comprises 14 questions assessing four domains of social cognition: theory of mind, emotional processes, attributional style and social knowledge. The score range from 28 to 140 points. The higher the score, the greater the impact of the disorders is considered.
  The questionnaire will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a daily life impact self-questionnaire 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  The ERF-CS (Echelle de Répercussion Fonctionnelle des troubles de la Cognition Sociale; Peyroux & Franck, 2014), administered to the participant, comprises 14 questions assessing four domains of social cognition: theory of mind, emotional processes, attributional style and social knowledge. The score range from 28 to 140 points.. The higher the score, the greater the impact of the disorders is considered.
  The questionnaire will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.
Change from a daily life impact hetero-questionnaire 48 hours after the end of the therapy | Baselines, 24-48 hours after the last session of the therapy
  The questionnaire (Taché, 2014), administered to someone close to the participant, includes 24 questions aimed at evaluating three areas of the theory of mind: social participation, conversation management and perspective taking. The score range from 24 to 96 points. The lower the score, the greater the impact of the disorders is considered.
  The questionnaire will be administered before the therapy (baselines) and directly (24-48 hours) after the last session of the therapy to analyze the change of performance.
Change from a daily life impact hetero-questionnaire 1 month after the end of the therapy | Baselines, 1 month-follow-up
  The questionnaire (Taché, 2014), administered to someone close to the participant, includes 24 questions aimed at evaluating three areas of the theory of mind: social participation, conversation management and perspective taking. The score range from 24 to 96 points. The lower the score, the greater the impact of the disorders is considered.
  The questionnaire will be administered before the therapy (baselines) and one month after the last session of the therapy to analyze the long-term change of performance.
Maintenance from a daily life impact hetero-questionnaire 1 month after the end of the therapy | 24-48 hours after the last session of the therapy, 1 month-follow-up
  The questionnaire (Taché, 2014), administered to someone close to the participant, includes 24 questions aimed at evaluating three areas of the theory of mind: social participation, conversation management and perspective taking. The score range from 24 to 96 points. The lower the score, the greater the impact of the disorders is considered.
  The questionnaire will be administered 24-48 hours and one month after the last session of the therapy to analyze the maintenance of performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Neuchâtel, Neuchâtel, Switzerland